CLINICAL TRIAL: NCT04772937
Title: Comparison of Two Surgical Approaches in the Treatment of Cervical Dysplasia: Complete Removal of the Transformation Zone (LLETZ) Versus Isolated Resection of the Colposcopically Visible Lesion (LEEP)
Brief Title: Comparison of LLETZ Versus LEEP for the Treatment of Cervical Dysplasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Clemens Tempfer, Principal Investigator, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LLETZ-2
Record Dates: First submitted 2021-02-22; First posted 2021-02-26 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Cervical Dysplasia
Keywords: cervical dysplasia; conization; surgery; cervical cancer; LLETZ; LEEP
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective randomization, 1:1 allocation, group 1: LLETZ, group 2: LEEP
Who Masked: Participant
Masking Description: Patient is anesthetized during surgery and will not recognize type of surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LLETZ group (Other): LLETZ (large loop excision of the transformation zone) is one of several possible surgical interventions for treating cervical dysplasia.
  Interventions: Procedure: LLETZ
- LEEP group (Other): LEEP (loop electrosurgical excision procedure) is one of several possible surgical interventions for treating cervical dysplasia.
  Interventions: Procedure: LEEP

INTERVENTIONS:
Procedure: LLETZ — LLETZ is one of several possible surgical interventions for treating cervical dysplasia. The transformation zone of the cervix is completely removed
  Other Names: Large Loop Excision of the Transformation Zone
  Arms: LLETZ group
Procedure: LEEP — LEEP is one of several possible surgical interventions for treating cervical dysplasia. Only the dysplastic lesion is removed without removing the whole transformation zone.
  Other Names: Loop Electrosurgical Excision Procedure
  Arms: LEEP group

SUMMARY:
Cervical dysplasia is the precursor of cervical cancer. LEEP and LLETZ are standard surgical procedures to treat cervical dysplasia. There is no direct head-to-head comparison between LEEP and LLETZ in the literature regarding oncologic safety, for which complete resection of the dysplastic lesion (so-called 'in-sano resection') is the most appropriate postoperative surrogate parameter. Further clinical studies are therefore useful to optimize surgical therapy for cervical dysplasia.

The primary objective of the present study is to compare LLETZ (resection of the dysplastic lesion including the transformation zone) with targeted resection of the colposcopically conspicuous lesion only (LEEP) and to compare it with regard to oncological safety (defined as non-in-sano rate).

DETAILED DESCRIPTION:
Cervical cancer is one of the most common cancers in women and one of the leading causes of death in women worldwide. Pre-cancerous lesions (dysplasias) are detected by the preventive smear test at the gynecologist and can thus contribute to a 100% chance of cure if they are clarified by a colposcopic examination as part of the dysplasia consultation and dysplastic lesions are then surgically removed if necessary (conization).

In practice, there are four different methods by which conization can be performed: Knife Conization, Laser Conization, Large Loop Excision of the Transformation Zone (LLETZ) and Loop Electrical Excision Procedure (LEEP). The first three methods have in common that they aim to remove the entire transformation zone. The rationale for this is that both the precancerous lesions and the cervical carcinoma itself originate in the transformation zone of the cervix. This thesis would support the idea of resecting the lesion while taking the remaining healthy transformation zone along as a precaution. However, it is clear that with the removal of the entire transformation zone, healthy tissue is removed in addition to the lesion itself. Any increase in radicality may increase the complication rate of the procedure, especially with regard to the most feared long-term complication of preterm birth, because the more cervical tissue is removed, the higher the risk of subsequent preterm birth. This connection speaks in favor of the use of LEEP, in which only the visible dysplastic tissue in healthy tissue is removed in the sense of a radical resection, without at the same time also removing the entire transformation zone, especially in women who still wish to have children.

In summary, the aim of conization is on the one hand to achieve a high level of oncological safety (low recurrence rate, high R0 resection rate) by resecting sufficient dysplastic tissue, and on the other hand to avoid excessive tissue resection, because this would increase the risk of premature birth in a subsequent pregnancy.

There is no direct head-to-head comparison between LEEP and LLETZ in the literature regarding oncologic safety, for which complete resection of the dysplastic lesion (so-called 'in-sano resection') is the most appropriate postoperative surrogate parameter. In a Pubmed literature search (search date: February 10, 2021, search terms: conization, LEEP, LLETZ, resection margin, randomized), no prospective randomized study on this topic was found. Further clinical studies are therefore useful to optimize surgical therapy for cervical dysplasia

The primary objective of the present study is to compare LLETZ (resection of the dysplastic lesion including the transformation zone) with targeted resection of the colposcopically conspicuous lesion only (LEEP) and to compare it with regard to oncological safety (defined as non-in-sano rate).

For this purpose, patients with histologically confirmed CIN II/III will be randomly assigned to one of the two surgical methods. In order to exclude an unwanted influence by unconsciously different behavior of the patients, the patient will only learn about the surgical method performed on her after the control examination 6 months postoperatively (unilateral blinding). The surgeon is not blinded for obvious technical reasons. However, in case of complications, access to the surgical report and the chosen method is possible at any time.

Immediately postoperatively, the specimen is examined histologically and evaluated with regard to the depth of the conus and the degree of dysplasia as well as the resection margins (R0= free resection margin; R1= dysplasia extends to the resection margin) by a pathology specialist.

After an interval of 6-8 months, the first follow-up examination (the so-called "test of cure") with PAP smear and HPV test is performed in accordance with the guidelines. The two groups are compared with regard to normalization of the Pap smear, HPV status and colposcopic findings (including histology in the case of colposcopic abnormalities).

For patients with negative HPV test, unremarkable cytology, histology and colposcopy, the study is terminated. These patients are considered cured and discharged to regular screening with their established gynecologist. In case of abnormalities, the further procedure is determined according to the usual clinical criteria in conformity with the guidelines: clinical control after 3 and/or 6 months or re-conization.

Secondary target criteria of the study are, in addition to the intra- and postoperative complication rate, the pain perception of the patients and the intraoperative blood loss, also the rate of negative high risk HPV tests after 6-8 months, since a negative HPV test is generally regarded as evidence of successful treatment. Thus, the negative predictive value for a negative HPV test after conization ranges from 92% to 100%. Successful therapy usually results in elimination of the HP virus. Accordingly, a negative HPV test excludes CIN persistence or recurrence with a high probability. In contrast, a persistently positive HPV test may be taken as an indication of persistence of dysplasia or as an indicator of recurrent dysplasia.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed High Grade Squamous Intraepithelial Lesion (HSIL)
* Colposcopically visible lesion
* No therapy of the disease so far

Exclusion Criteria:

* Pregnancy of the patient at/after inclusion in the study; pregnancy after conization and before the control after 6 months is possible and does not lead to exclusion from the study.
* Taking immunosuppressive drugs (incl. glucocorticoids)
* Known HIV positivity
* Malignant disease requiring treatment
* Unsatisfactory colposcopy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Surgical specimen margin status | Pathology assessment of the cone specimen (within 2-4 days after surgery)
  Oncological safety as defined by the rate of specimens with involved margins, i.e. cervical dysplasia present at the edge of the surgical specimen.

SECONDARY OUTCOMES:
Intraoperative and postoperative complication rate | During and within 3 weeks after the procedure
  Rate of complications such as excessive bleeding, re-operation, unplanned readmission, infection
Cone size | During surgery
  Size of the resected tissue
Patient's pain | Immediately after the surgery
  Pain experienced by the patients (11-item Visual Analogue Scale); minimum 0 (no pain), maximum 10 (unbearable pain)
HPV clearance | 6 months post surgery
  HPV high-risk positivity by PCR
Cone volume | During surgery
  Volume of the resected tissue

CONTACTS AND LOCATIONS:
Overall Officials: Clemens B Tempfer, MD, MBA, Principal Investigator — Ruhr-Universität Bochum / Marien Hospital Herne
Locations (1):
- Dept. OBGYN Ruhr University Bochum, Herne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin-Hirsch PP, Paraskevaidis E, Bryant A, Dickinson HO. Surgery for cervical intraepithelial neoplasia. Cochrane Database Syst Rev. 2013 Dec 4;2013(12):CD001318. doi: 10.1002/14651858.CD001318.pub3. PMID 24302546
- [Background] Chua KL, Hjerpe A. Human papillomavirus analysis as a prognostic marker following conization of the cervix uteri. Gynecol Oncol. 1997 Jul;66(1):108-13. doi: 10.1006/gyno.1997.4753. PMID 9234930